CLINICAL TRIAL: NCT02142426
Title: A Retrospective Analysis of Laboratory Testing on Chronic Wound Patients
Status: Completed | Type: Observational
Sponsor: Southwest Regional Wound Care Center (Other)
Responsible Party: Principal Investigator, Randall Wolcott, Prinicipal Investigator, Southwest Regional Wound Care Center
Other Study IDs: 56-RW-021
Record Dates: First submitted 2011-09-13; First posted 2014-05-20 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Wound Chronic Draining
Keywords: wound chronic

STUDY DESIGN:
Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — To pursue statistical analysis on a series of molecular laboratory results obtained from chronic wounds
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study was to pursue statistical analysis on a series of molecular laboratory results obtained from chronic wounds. It elucidated diversity, quantification, and other aspects of microbial diversity in chronic wounds.

DETAILED DESCRIPTION:
The information was processed from culture results that were processed to compile an antibiogram for a laboratory.

ELIGIBILITY:
Inclusion Criteria:

-Patients with chronic wounds.

Exclusion Criteria:

-Patients without chronic wounds.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronic wound patients
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Improve selection of systemic antibiotics based on results using molecular diagnostics. | 1 year
  The study elucidated diversity, quantification, and other aspects of microbial diversity in chronic wounds. It evaluated samples from different regions, different types of wounds, different outcomes, and longitudinal data if multiple samples were sent over time from a single individual.

SECONDARY OUTCOMES:
2. Data Collection: The molecular wound cultures have been performed on thousands of patients from around the country. The information from the culture results that were processed were used to compile an antibiogram for a laboratory. | 1 year
  There are many geographic regions which have a number of samples which could be analyzed and compared to other geographic regions yielding valuable insight into the microbiology of chronic wounds.

CONTACTS AND LOCATIONS:
Overall Officials: Randall D Wolcott, MD, Principal Investigator — Southwest Regional Wound Care Center
Locations (1):
- Southwest Regional Wound Care Center, Lubbock, Texas, United States

REFERENCES:
- [Result] Dowd SE, Wolcott RD, Kennedy J, Jones C, Cox SB. Molecular diagnostics and personalised medicine in wound care: assessment of outcomes. J Wound Care. 2011 May;20(5):232, 234-9. doi: 10.12968/jowc.2011.20.5.232. PMID 21647068